CLINICAL TRIAL: NCT02327611
Title: CUstodiol Versus RInger: whaT Is the Best Agent? A Randomized Double Blind Trial.
Brief Title: CUstodiol Versus RInger: whaT Is the Best Agent?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, yamume tshomba, Medical Doctor Associate Professor of Vascular Surgery, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CURITIBA/9/OSR
Record Dates: First submitted 2014-12-15; First posted 2014-12-30 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Thoracoabdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Custodiol (Experimental): Renal perfusion with Custodiol (cold crystalloid solution enriched with histidine-tryptophan-ketoglutarate).
  Interventions: Drug: Custodiol
- enriched Ringer's lactate solution (Active Comparator): Renal perfusion with cold Ringer's lactate solution enriched with methylprednisolone 125 mg /L and mannitol 12.5 g /L.
  Interventions: Drug: Enriched Ringer's lactate solution

INTERVENTIONS:
Drug: Custodiol
  Arms: Custodiol
Drug: Enriched Ringer's lactate solution
  Arms: enriched Ringer's lactate solution

SUMMARY:
Postoperative renal failure is the most significant risk factor for early mortality after elective surgical repair of thoracoabdominal aortic aneurysms (TAAAs).

To prevent damages related to kidney ischemia during aortic crossclamping and TAAA repair, the most recent guidelines recommend the use of cold crystalloid or blood perfusion. Since the most studied crystalloid solution is the Ringer's lactate solution, this can be considered the standard of care for evaluating the effectiveness of other substrates.

An histidine-tryptophan-ketoglutarate enriched crystalloid solution named Custodiol (Dr. Franz Kohler Chemie GmbH, Bensheim, Germany) is currently used for organ preservation during transplantation and for cardioplegia during open-heart surgery in most EU countries. This solution may provide a better grade of renal protection to ischemic damage than the standard crystalloid solutions.

A recent observational study published by our group suggested a lower incidence of postoperative renal kidney injury in patients undergoing open TAAA surgical repair using renal perfusion with Custodiol, as compared to those perfused with an enriched Ringer's lactate solution.

Objective of this study is the confirmation of the promising findings about the effectiveness of renal perfusion with Custodiol during repair of TAAA compared with other crystalloid.

The study will be a prospective, single-center, randomized, double-blind, controlled trial, investigating Acute Kidney Injury in patients undergoing TAAA open repair using Custodiol renal perfusion versus an enriched Ringer's lactate solution. It is expected to enroll adult patients undergoing elective TAAA open repair. Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Ability to provide written informed consent; Patient undergoing open surgical repair of TAAA requiring renal perfusion.

Exclusion Criteria:

1. Patients who have participated to experimental trials during the previous 3 months
2. Intervention under emergency / urgency
3. Patient uncooperative and / or affected by mental disease
4. Allergy or intolerance to the study drug
5. Patient under renal replacement treatment (dialysis) before surgery
6. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | Kidney function will be assessed during hospital stay (an expected average of 2 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy